CLINICAL TRIAL: NCT04153994
Title: Pediatric Scoliosis Surgery: Enhanced Recovery With Erector Spinae Plane Blockade Utilizing Surgically Placed Catheters
Brief Title: Erector Spinae Plane Blockade in Pediatric Scoliosis Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52852
Record Dates: First submitted 2019-10-24; First posted 2019-11-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Scoliosis; Juvenile; Scoliosis; Adolescence
Keywords: Erector Spinae Plane Blockade; Pediatric Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Blockade Treatment (Experimental): Patients will receive an erector spinae plane blockade prior to their surgery as per standard regional anesthesia technique.
  Interventions: Procedure: Erector Spinae Plane Blockade
- Erector Spinae Plane Blockade Control - Standard of Care (No Intervention): Patients will receive the standard of care for pediatric scoliosis surgery including multi-modal opioid pain management. If the patient declines to consent to enrollment into the randomized study, patients may still participate by allowing prospective data and samples collection/analysis with respect to perioperative choice.

INTERVENTIONS:
Procedure: Erector Spinae Plane Blockade — The ESPB is fascial plane block performed by injecting local anesthetic between the erector spinae muscle and the transverse process. Its proposed mechanism of action is via blockade of the dorsal and ventral rami of the thoracic spinal nerves and sympathetic fibers.
  Arms: Erector Spinae Plane Blockade Treatment

SUMMARY:
Providing effective analgesia after spinal fusion for idiopathic scoliosis remains a challenge with significant practice variation existing among high volume spine surgery centers. Even in the era of multimodal analgesia, opioids are the primary analgesics used for pain control after pediatric scoliosis surgery, but have multiple known adverse effects. The erector spinae plane block (ESPB) is a newly described fascial plane block performed by injecting local anesthetic between the erector spinae muscle and the transverse process. Additionally, there are case reports describing the ESPB as part of a multi-modal analgesic plan in adult degenerative spine surgery as well as adult spinal deformity surgery, demonstrating effective analgesia and no clinical motor blockade. Although it is known that the inflammatory reaction plays a crucial role in the mechanism of acute pain after major surgery, the effectiveness of the current regional approach on inflammatory response is not well studied.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Diagnosed with Idiopathic scoliosis
* Undergoing single-stage posterior spinal instrumentation and fusion

Exclusion Criteria:

* Thorascopic tethering procedure
* Two-stage procedure
* Abnormal developmental profile
* Congenital/neuromuscular scoliosis
* Requiring PICU admission
* Known allergy to lidocaine
* Known cardiac, renal or liver disease or dysfunction
* Pre-existing pain complaints, i.e. on regular analgesic medications
* Current psychiatric diagnosis, e.g. anxiety, depression, eating disorder, defined according to DSM criteria.
* Requiring non-standard post-op pain management
* Any history of seizures
* Unplanned staged procedure
* Weight < 5th centile or > 85th centile for age
* Porphyria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Length of Stay (LOS) | Through hospital stay, an average of 5 days
  Determine if bilateral surgical placed ESPBs will decrease length of stay in the pediatric ICU and the hospital. LOS and decrease postoperative opioid consumption.)
Postoperative Opioid Consumption | Through hospital stay, an average of 5 days
  Determine if bilateral surgical placed ESPBs will decrease postoperative opioid consumption measured in Morphine Milligram Equivalents (MME)
Maximum lidocaine plasma concentration [Cmax] | Through hospital stay, an average of 5 days
  Measure daily serial plasma lidocaine levels from ESPB catheters
Patient-Reported Pain Scores | Through hospital stay, an average of 5 days
  Patients will be asked on a daily basis by the research staff to report pain scores on a scale of 1-10 (1 signifying no pain to 10 signifying the worse pain).
Inpatient Postoperative Mobility | Through hospital stay, an average of 5 days
  Inpatient postoperative mobility will be tracked using activity tracker accelerometers and subsequently compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Sheffer BW, Kelly DM, Rhodes LN, Sawyer JR. Perioperative Pain Management in Pediatric Spine Surgery. Orthop Clin North Am. 2017 Oct;48(4):481-486. doi: 10.1016/j.ocl.2017.06.004. Epub 2017 Jul 15. PMID 28870307
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kose HC, Kose SG, Thomas DT. Lumbar versus thoracic erector spinae plane block: Similar nomenclature, different mechanism of action. J Clin Anesth. 2018 Aug;48:1. doi: 10.1016/j.jclinane.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29649625
- [Background] Almeida CR, Oliveira AR, Cunha P. Continuous Bilateral Erector of Spine Plane Block at T8 for Extensive Lumbar Spine Fusion Surgery: Case Report. Pain Pract. 2019 Jun;19(5):536-540. doi: 10.1111/papr.12774. Epub 2019 Mar 15. PMID 30758122
- [Background] Kline J, Chin KJ. Modified dual-injection lumbar erector spine plane (ESP) block for opioid-free anesthesia in multilevel lumbar laminectomy. Korean J Anesthesiol. 2019 Apr;72(2):188-190. doi: 10.4097/kja.d.18.00289. Epub 2018 Nov 2. No abstract available. PMID 30392347
- [Background] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Background] Demmy TL, Nwogu C, Solan P, Yendamuri S, Wilding G, DeLeon O. Chest tube-delivered bupivacaine improves pain and decreases opioid use after thoracoscopy. Ann Thorac Surg. 2009 Apr;87(4):1040-6; discussion 1046-7. doi: 10.1016/j.athoracsur.2008.12.099. PMID 19324125